CLINICAL TRIAL: NCT02519478
Title: Prevention of Head Impacts in Football: The HuTT Technique
Acronym: HuTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Hampshire (Other)
Collaborators: University of Michigan (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Erik Swartz, Professor, University of New Hampshire
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UNH-02-5779-01
Record Dates: First submitted 2015-08-04; First posted 2015-08-11 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Head Trauma; Cognitive Manifestations
Keywords: football; Training Techniques; education; Athletic Injuries; Brain Concussion
MeSH Terms: conditions — Craniocerebral Trauma; Neurobehavioral Manifestations; Athletic Injuries; Brain Concussion

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Helmetless Tackling Training (HuTT) (Experimental): The HuTT program is modeled after a tackling drill progression common to the sports of rugby and American football, but participants do not wear helmets or should pads as they normally would in football. Drills will be executed at 50%-75% effort. The goal of the contact is to execute proper technique. Drills will be supervised at all times and feedback will be provided to confirm proper technique and correct improper technique. The HuTT drill will be completed in two phases and takes approximately 6-10 minutes per session. A research assistant will ensure adherence and standardization of the treatment throughout the season. Subjects in the intervention group will participate in HuTT 4 times per week throughout the 2 weeks of pre-season and 2 times a week during in-season.
  Interventions: Behavioral: Helmetless Tackling Training (HuTT)
- Control (No Intervention): Control group subjects participate in normal football activities as they would normally have during a football season

INTERVENTIONS:
Behavioral: Helmetless Tackling Training (HuTT) — see previous sections
  Arms: Helmetless Tackling Training (HuTT)

SUMMARY:
The purpose of the study is to determine the effectiveness of the helmet-less tackling training (the HuTT Technique) intervention to reduce head impacts in high school football players and to gain an understanding of the neurocognitive effects of repetitive head impacts in football. The investigators hypothesis is that the HuTT Technique will result in a reduced frequency and magnitude of helmet impacts than the control group measured by a head impact measurement system. Also, the investigators hypothesize the HuTT Technique group will demonstrate less changes in neurocognitive scores in the mid and post season evaluations compared to the control group. Head impacts will be measured using the SIM-G impact monitor made by Triax Technology. The SIM-G impact monitor measures the location, magnitude, and direction of every head impact in real time and is stored on a protected cloud-based system. The sensor is worn by each athlete in a headband or skullcap. Neurocognitive function will be measured using the Immediate Post-concussion Assessment and Cognitive Testing (ImPACT) test. The test is used as a tool to determine baseline neurocognitive function and is used in comparison if an athlete was to be injured to ensure he/she returns to baseline. ImPACT measures memory (verbal, visual, working), processing speed and reaction time using a variety of tests. Subjects will be recruited from local high school football teams and will include freshman, sophomores and juniors. Since the study is expected to run for 2 years, seniors will not be eligible for participation. The target is to recruit at least 150 total subjects. All subjects will be equipped with a new helmet that is fitted to their head and a headband that will be used to hold the head impact telemetry sensor. In addition, all subjects will take an ImPACT test preseason, midseason and postseason. At the conclusion of each season, all of the impacts from the SIM-G impact monitor system and ImPACT test scores will be analyzed. The relevant outcome measures to be analyzed include head impact frequency, location, magnitude, symptom scores, memory, visual motor speed and reaction time composite scores. Statistical analysis will be used to determine if the HuTT intervention minimized head impacts and neurocognitive decline compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* high school football participant
* two years eligibility

Exclusion Criteria:

* one year eligibility (high school senior)
* use of a Riddell Speed "Flex" helmet

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Head(helmet) Impact frequency | Participants will be followed for the duration of the football season, an expected average of 11 weeks
  The number of times a football participant sustains and impact to their helmet during practices or games, except 'walk-throughs' for two seasons.
Change in Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT) computerized concussion evaluation system Test Scores | Change from baseline scores at an average of 6 weeks and 11 weeks
  A sophisticated computerized neuropsychological performance test for cognitive performance

SECONDARY OUTCOMES:
Head(helmet) Impact magnitude | Participants will be followed for the duration of the football season, an expected average of 11 weeks
  The acceleration of force from an impact a football participant sustains to their helmet during practices or games, except 'walk-throughs' for two seasons.
Head(helmet) Impact location | Participants will be followed for the duration of the football season, an expected average of 11 weeks
  The location of the impacts a football participant sustains during practices or games, except 'walk-throughs' for two seasons.
Head(helmet) Impact duration | Participants will be followed for the duration of the football season, an expected average of 11 weeks
  The duration (milliseconds) of the impacts a football participant sustains during practices or games, except 'walk-throughs' for two seasons.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Swartz, PhD, Principal Investigator — University of New Hampshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Swartz EE, Myers JL, Cook SB, Guskiewicz KM, Ferrara MS, Cantu RC, Chang H, Broglio SP. A helmetless-tackling intervention in American football for decreasing head impact exposure: A randomized controlled trial. J Sci Med Sport. 2019 Oct;22(10):1102-1107. doi: 10.1016/j.jsams.2019.05.018. Epub 2019 Jun 7. PMID 31204104
- See also: Announcement of award to fund study with video of feasibility study being conducted at organization — https://ninesights.ninesigma.com/web/head-health/awardees